CLINICAL TRIAL: NCT05003284
Title: Effect of Acupressure Application on Patients' Nausea, Vomiting, Pain, and Sleep Quality After Laparoscopic Cholecystectomy: A Randomized Placebo-controlled Study
Brief Title: Effect of Acupressure Application on Patients' Nausea, Vomiting, Pain, and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tülay KILINÇ, Principal İnvestigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: tulay25
Record Dates: First submitted 2021-06-25; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Complications
Keywords: acupressure; nausea-vomiting; nurse; pain; PC6; sleep
MeSH Terms: conditions — Postoperative Complications; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure wristband (Experimental): On the day before the surgery, the patients in the experimental groups were introduced to the wristband and given an explanation regarding how it should be used. Approximately 30 minutes before the experimental group patients went to surgery, the PC6 acupressure point was determined for the patients. Immediately after the experimental group patients were taken to the wards after surgery, wristbands were placed on both wrists. İt was stated to the patients that the wristbands should remain on for 24 hours. The wristband was removed at the end of the 24th hour.
  Interventions: Device: acupressure wristband
- placebo wristband (Placebo Comparator): On the day before the surgery, the patients in the placebo groups were introduced to the wristband and given an explanation regarding how it should be used. Approximately 30 minutes before the placebo group patients went to surgery, the PC6 acupressure point was determined for the patients. Right after their surgery, patients in the placebo group were fitted with a wristband that looked the same as the acupressure wristband but did not have an acupressure application head. İt was stated to the patients that the wristbands should remain on for 24 hours. The wristband was removed at the end of the 24th hour.
  Interventions: Device: placebo wristband

INTERVENTIONS:
Device: acupressure wristband — acupressure after surgery
  Arms: acupressure wristband
Device: placebo wristband — acupressure after surgery
  Arms: placebo wristband

SUMMARY:
This study was conducted to determine the effect of acupressure on nausea, vomiting, pain, and sleep quality after laparoscopic cholecystectomy. This was a randomized controlled experimental study with a placebo group. The sample comprised 188 patients who underwent laparoscopic cholecystectomy (control:64; experimental:64; and placebo:60). Acupressure was performed on the experimental and placebo groups with a wristband for 24 hours.

DETAILED DESCRIPTION:
Despite scientific developments and the antiemetic and analgesic drugs used, postoperative nausea, vomiting, and pain continue to be major problems affecting patients today. Many different pharmacological approaches have been developed to minimize postoperative nausea, vomiting, and pain. However, the side effects associated with traditional antiemetics and analgesics and the high cost of drugs have resulted in an increase in the use of non-pharmacological methods. Acupressure, one of such non-pharmacological methods, is based in traditional Chinese medicine. It is a treatment method that ensures proper functioning of energy channels through the application of pressure to the acupressure points on the meridians carrying energy in the body using palms, fingers, or special stimulation bands. Acupressure is an application included in the classification of nursing interventions. In the classification of nursing interventions, it is stated that acupressure is effective in relief, reduction of pain, elimination and prevention of nausea, and it is recommended to be applied to patients. Acupressure supports the independent role of nurses and provides evidence-based practice for nurses in symptom management.

Acupressure is a noninvasive, easy-to-apply, safe, low-cost application with no side effects. Thus, it is a complementary alternative treatment method that is increasingly used in the prophylaxis and treatment of postoperative nausea and vomiting due to the absence of drug-related side effects and pain and better tolerability in patients. Most of the non-pharmacological studies on the reduction of nausea and vomiting focus on the stimulation of the Pericardium 6 (PC6) acupressure point at the wrist. The nervous system is activated by the stimulation of the PC6 point on the pericardium meridian, and this system sends signals to the brain, which results in an antiemetic effect. After the brain is stimulated, neurotransmitters such as serotonin, dopamine, and endorphins are secreted. These substances prevent nausea and vomiting by blocking chemicals that can cause nausea. Acupressure is also a frequently used non-pharmacological method for reducing pain and regulating sleep. The endorphins and serotonin secreted by the stimulation of acupressure points create a calming response in the body, reduce anxiety, induce relaxation, and improve sleep quality. In addition, acupressure stimulation regulates parasympathetic nervous system activity. This situation increases sleep quality by providing an increase in autonomous responses and a decrease in psychological stress.

This study was conducted to determine the effect of acupressure on nausea, vomiting, pain, and sleep quality after laparoscopic cholecystectomy. This was a randomized controlled experimental study with a placebo group. The sample comprised 188 patients who underwent laparoscopic cholecystectomy (control:64; experimental:64; and placebo:60).

IMPACT STATEMENT What is already known on this subject? Nausea, vomiting, pain and insomnia in the postoperative period may cause discomfort, and this may adversely affect the patient's compliance with the treatment. Managing nausea, vomiting and pain in the postoperative period and improving the quality of sleep are among the important responsibilities of nurses. Thus, acupressure, as a complementary alternative method, can be recommended to reduce nausea and vomiting and improve sleep quality after surgical intervention. Acupressure is effective in relief, reduction of pain, and relief and prevention of nausea and vomiting. Acupressure supports the independent roles of nurses, provides evidence-based practice to nurses in symptom management, and improves patient-nurse relationships.

What the implications are of these findings for clinical practice and/or further research? This study is important because it shows that acupressure can be used as a complementary and alternative method in the postoperative period. Although it is reported that acupressure, which is a safe and effective method, can reduce the rate of complications, increase patient comfort, and thus affect the success of the surgical process when applied before or after surgical intervention, more evidence-based studies are needed to clearly demonstrate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 65 years,
* Underwent laparoscopic cholecystectomy under general anesthesia,
* Conscious, were able to communicate, had no hearing or speech problems,
* Volunteered to participate were included in the study.

Exclusion Criteria:

* Patients who left the study at any stage,
* Taken to the intensive care unit in the early postoperative period, or underwent extra surgical interventions (e.g., hernia repair, etc.) were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Numeric nausea scale. | up to 24 hours
  The numeric nausea scale is a self-reported scale from 0 to 10, with 0 indicating "no nausea" and 10 indicating "very severe nausea" The highest nausea severity felt by the patient is marked on the scale
Visual analog scale | up to 24 hours
  The visual analog scale was used to evaluate the pain severity of the patient. It is a self-reported scale in the form of a 10-cm ruler indicating no pain at one end and unbearable pain at the other. Accordingly, the patient is told to evaluate his/her pain between 0 and 10, with 0 indicating "no pain" and 10 indicating "unbearable pain
Verbal category scale. | up to 24 hours
  The verbal category scale is a one-dimensional, simple, descriptive scale. Patients are asked to state the most appropriate word to describe their pain while filling in the scale. To describe the severity of pain, the patients had to choose from among (1) mild, (2) disturbing, (3) severe, (4) very severe, and (5) unbearable
Richards-Campbell Sleep Questionnaire | To collect data on sleep, richards-campbell sleep questionnaire was applied to all three groups 24 hours after surgery to evaluate sleep, and the responses were recorded
  Richards-campbell sleep questionnaire evaluates the depth of night sleep, sleep latency, number of awakenings, return to sleep, sleep quality, and the level of noise in the environment. It consists of six questions in total. Each item of the scale is evaluated with a visual analog scale ranging from 0 to 100. In this scale, "0-25" points indicate "very poor sleep" and "76-100" points indicate "very good sleep."

CONTACTS AND LOCATIONS:
Overall Officials: Tülay kılınç, Dr, Principal Investigator — Ataturk Unıversty
Locations (1):
- Tülay Kılınç, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No